CLINICAL TRIAL: NCT06945471
Title: Impact of Computer-Mediated Versus Face-to-Face Motivational-Type Interviews on Participants' Language and Subsequent Cannabis Use: Randomized Controlled Trial
Brief Title: Computer-Mediated Versus Face-to-Face Motivational-Type Interviews
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 219115-2; 5R24DA029989-05 (NIH)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Marijuana Use
Keywords: Motivational interviews; computer-mediated; commitment language; change talk; marijuana use; randomized study; young adults
MeSH Terms: conditions — Marijuana Use

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two conditions: 1) Face-to-face motivational type interviews or 2) Computer-mediated motivational type interviews.
Who Masked: Outcomes Assessor
Masking Description: We masked a participant's experimental condition (face-to-face motivational type interviews and computer-mediated motivational type interviews) when coding each interview, and thus minimized bias when evaluating the presence of commitment language within each interview transcript.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face motivational type (FTF MTIs) interviews (Experimental): The interviews conducted in this study were guided by 4 of the 5 major principles of MI. Specifically, the interviews (1) were nonjudgmental, (2) were empathic, (3) respected participants' autonomy, and (4) helped participants explore their ambivalence toward behavior change. However, unlike standard motivational interviews, the interviews in this study did not subtly guide participants toward reducing marijuana use. The interviews were not intended as a clinical intervention. The decision to omit the direction-oriented component of MI was guided by a single consideration: the national trend toward the legalization of recreational marijuana use. FTF MTIs were guided by a 4-page script that incorporated the main principles of MI, including reflective listening, expression of empathy, and a nonjudgmental conversational style. The script included an equal number of open-ended questions exploring the benefits and costs of using marijuana. FTF MTIs were conducted in a research office.
  Interventions: Behavioral: 1) Face-to-face, and 2) Computer-mediated motivational type interviews
- Computer-mediated motivational type interviews (CM-MTIs) (Experimental): Computer-mediated interviews were conducted using the identical 4-page script that guided the FTF MTIs. Computer-mediated MTIs were completed via computer, with the interviewer and participant located in adjacent rooms within the same research suite used for the FTF MTIs. However, the interviewer and interviewee never met in person. Upon arrival, a research assistant greeted participants, administered Time 1 assessments, and provided instructions for using the computer's instant messaging software to communicate during the motivational-type interview. LAN Instant Messenger software (version 1.2.35, Qualia Digital Solutions) was used to conduct computer-mediated interviews and computer-mediated MTIs were saved as text files.
  Interventions: Behavioral: 1) Face-to-face, and 2) Computer-mediated motivational type interviews

INTERVENTIONS:
Behavioral: 1) Face-to-face, and 2) Computer-mediated motivational type interviews

SUMMARY:
This study looks at whether in-person and computer-based motivational type interviews lead to the same kind of language and behavior change in young adults when they talk about their marijuana use. Researchers compared how much participants talked about wanting to change their level of marijuana use (change talk) or maintain their level of marijuana use (sustain talk) during each type of interview. Researchers investigated if change talk and sustain talk predicted who continued to use or not use marijuana. All participants completed:

* A survey assessing their frequency of marijuana use.
* A brief motivational type interview, either a face-to-face-motivational type interview or computer-mediated motivational type interview.
* A two-month follow-up survey, again assessing their level of marijuana use.

DETAILED DESCRIPTION:
This study investigated if face-to-face motivational-type interviews (FTF-MTIs) and computer-mediated MTIs elicit the same amount of "change talk" and behavior change when young adults discuss their ambivalence about using marijuana. 150 young adults participated in the study: 50 frequent marijuana users, 50 occasional marijuana users, and 50 non-marijuana users. All participants reported being at least moderately ambivalent about their current level of marijuana use. Participants were randomly assigned to complete a brief MTI using either the standard face-to-face format or a computer-mediated format. Amrhein's manual for assessing the presence of "change talk" and "sustain talk" was used to code the language produced by respondents in each interview format. Participants' level of marijuana use was assessed at a 2-month follow-up. We hypothesized the following:

* FTF MTIs would elicit more words than computer-mediated MTIs
* FTF MTIs would take less time to complete than compute-mediated MTIs.
* Participants who used language denoting a strong commitment to reduce their marijuana use would report significantly less marijuana use at the 2-month follow-up compared with participants whose MI-type interviews contained weaker commitment language, regardless of interview format (FTF or computer-mediated).
* FTF MTIs and computer-mediated MTIs would elicit the same amount of sustain talk and change talk (e.g., desire, ability, reasons, need, commitment, and readiness statements). The latter hypothesis was exploratory because no previous research has compared these two formats for conducting MTIs.

ELIGIBILITY:
Inclusion Criteria:

* A brief eligibility questionnaire assessed each respondent's age, previous marijuana use, and ambivalence about their marijuana use during the year preceding the study. Sample ambivalence items included: "During the past year I've had mixed emotions about my level of marijuana use or nonuse," and "How much have you thought about changing your marijuana use or nonuse during the past year?" Responses options ranged from 0 ("not at all") to 5 ("medium amount") to 10 ("a lot"). Respondents who were 18-29 years of age and reported at least a "medium amount" of ambivalence in response to 2 or more ambivalence questions were eligible to participate in the study. Three types of adults were recruited: non-marijuana users, occasional marijuana users, and frequent marijuana users. Non-marijuana users were defined as individuals who reported no history of marijuana use in their lifetime. Occasional marijuana users were defined as individuals who used marijuana 1-5 times during the 2 months preceding the study but fewer than 24 times during the year preceding the study. Frequent marijuana users were defined as individuals who used marijuana more than 7 times during the 2 months preceding the study and more than 24 times during the year preceding the study.

Exclusion Criteria:

* We excluded participants who did not meet the above criteria.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Frequency of marijuana use at two-month follow-up | 2-month-follow-up
  During the past two months, how many times (if any) have you smoked or consumed marijuana?

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence D. Cohn, PhD, Principal Investigator — University of Texas, El Paso; Jon Amastae, PhD, Principal Investigator — University of Texas, El Paso
Locations (1):
- University of Texas at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated or analyzed during this study are available from the corresponding author on reasonable request. No individual raw data will be released that would compromise the anonymity or confidentiality of the participants.

REFERENCES:
- [Derived] Llanes KD, Amastae J, Amrhein PC, Lisha N, Arteaga K, Lopez E, Moran RA, Cohn LD. Impact of Computer-Mediated Versus Face-to-Face Motivational-Type Interviews on Participants' Language and Subsequent Cannabis Use: Randomized Controlled Trial. J Med Internet Res. 2025 Apr 25;27:e59085. doi: 10.2196/59085. PMID 40279644